CLINICAL TRIAL: NCT04300400
Title: Development of a Flowchart Reflecting the Current Attitude and Approach Towards the Idiopathic Overactive Bladder Treatment in Belgium: A Delphi Study
Brief Title: Treatment of the Overactive Bladder Syndrome: A Delphi Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Astellas Pharma Inc (Industry); Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: B670201835542
Record Dates: First submitted 2020-02-07; First posted 2020-03-09 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Overactive Bladder Syndrome
Keywords: Overactive bladder Syndrome; Delphi study; Treatment algorithm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Delphi panel: Urologists of the Belgian Working group of Functional Urology willing to participate on the Delphi project.
  Interventions: Other: Delphi questionnaire

INTERVENTIONS:
Other: Delphi questionnaire — Statements on OAB topics, rated along their level of appropriateness on a scale from 1 to 9. Multiple rounds are organised to reach consensus on a topic.

SUMMARY:
Idiopathic overactive bladder syndrome (iOAB) is a prevalent condition in urological practice. The variability in management between specialists and between centers remains high. Even guidelines are not always clear on the treatment management of drug therapy resistant OAB. Standardization in OAB treatment is needed.

DETAILED DESCRIPTION:
Guidelines on the overactive bladder syndrome (European Association of Urology, American Urology Association and International Consultation on Incontinence) are comparable but remain vague mainly on the level between conservative and major surgery. They do not specify combinations of medications and do not distinguish between intradetrusor botulinum toxin injections (BTX) and sacral neuromodulation (SNM) because of lack of evidence.

To reduce the variability in the treatment management of OAB, standardization is needed.

By use of a Delphi technique, the current perception of Belgian urologists towards the most appropriate treatment approach for idiopathic OAB (iOAB) was explored.

Based on these results a practical treatment algorithm for its use in daily clinical practice could be developed.

ELIGIBILITY:
Inclusion Criteria:

* Profession: MD, Urologist
* Member of the working group of Functional Urology

Exclusion Criteria:

* Retirement
* Non-operative as an urologist.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Belgian Urologists: members of the working group of Functional Urology.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Degree of consensus on the level of appropriateness | 8 months
  No consensus, trend towards consensus or consensus

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Ghijselings, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No